CLINICAL TRIAL: NCT03621709
Title: Multicenter Ambispective Study of Clinical Outcomes of the CoreValve™Evolut R™ 34mm System: All Comers Post-market Registry
Brief Title: CoreValve™ Evolut R™ 34 mm System Registry (CoreValve34)
Acronym: TAVI34mm
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Responsible Party: Sponsor
Other Study IDs: ACUN-VALV-001
Record Dates: First submitted 2018-05-25; First posted 2018-08-08 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Aortic Valve Stenosis; Transcatheter Aortic Valve Implantation
Keywords: TAVR; TAVI; Aortic valve stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CoreValve™ Evolut R™ 34mm: All consecutive real-world patients with aortic stenosis selected for TAVI as part of routine clinical care, using a CoreValve™ Evolut R™ 34mm during the inclusion period will be entered the registry.

SUMMARY:
With the introduction of the CoreValve™ Evolut R™ 34mm (Medtronic™) prosthesis, patients with severe symptomatic aortic stenosis (AS) and large aortic annulus have become eligible for transcatheter aortic valve implantation (TAVI). The aim of this study is to detect the number of TAVI candidates with large aortic annulus, and to evaluate the feasibility, efficacy, and safety of TAVI using the CoreValve™ Evolut R™ 34mm.

DETAILED DESCRIPTION:
With the current transcatheter valves available in the market, is possible to cover a wide range of patients with diverse and complex anatomies. Nevertheless, there is a subgroup of patient with large aortic annulus (diameter > 27 mm), in whom the implant of a transcatheter valve is not possible because there is no valve suitable for such as aortic annulus size.

With the introduction of the CoreValveTM EvolutionTM R 34mm, patients with an aorttic annulus dimension up to 29 mm in diameter have become eligible for TAVI. However, there is a lack of information regarding the number of patient with AS and this particular anatomy of the aortic annulus. Italian and Dutch registries have reported a prevalence between 6.5 to 12.3% with large aortic annulus requiring the previous CoreValveTM 31mm. Yet, there is no reported data regarding this population of patients in Spain. Also, the clinical use of this larger prosthesis covers a wider range of aortic rings and may enchance the procedural challenges, such as a little margin for proper valve placement, more likelihood of interference with mitral valve function and damage to the cardiac conduction system during the prosthesis deployment.

So far, no studies regarding clinical experiences with the CoreValveTM EvolutionTM R 34mm have been published. The scarce information currently available with this new device may be distant from those found in its daily clinical use in non-selected patients. The results of this Spanish nationwide registry will help to answer a scientific need of information regarding acute procedural results and mid

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years of age.
* Subject accepted participate and signed informed consent.
* Subject with severe symptomatic AS patients selected for TAVI by the Heart Team of each participating hospital.
* Patients anatomically suitable for the implantation of a CoreValve™ Evolut R™ 34mm with the approved indications by any feasible and appropriate vascular routes.
* Subject must agree to undergo all follow-up visits

Exclusion Criteria:

* High probability of non-adherence to the follow-up requirements.
* Explicit refusal of participation in the registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with severe symptomatic aortic stenosis undergo TAVI using the CoreValve™ Evolut R™ 34 mm will be included
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Safety: Stroke | 12 months
  Stroke (disabling), dichotomous qualitative variable: yes/no
Efficacy: prosthetic regurgitation at early post TAVI | 12 months
  Percent of subjects with ≤ mild prosthetic regurgitation at early post-implant (mild, Moderate or Severe)
Safety:Incidence of permanent pacemaker implant rate | 12 months
  Incidence of permanent pacemaker implant rate, dichotomous qualitative variable: yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Victor A Jiménez Díaz, MD, MPH, Principal Investigator — Hospital Álvaro Cunqueiro; Pablo Jiménez Díaz, MD, MPH, Study Director — Hospital Álvaro Cunqueiro
Locations (1):
- Hospital Alvaro Cunqueiro, Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Freeman RV, Otto CM. Spectrum of calcific aortic valve disease: pathogenesis, disease progression, and treatment strategies. Circulation. 2005 Jun 21;111(24):3316-26. doi: 10.1161/CIRCULATIONAHA.104.486738. No abstract available. PMID 15967862
- [Background] Osnabrugge RL, Mylotte D, Head SJ, Van Mieghem NM, Nkomo VT, LeReun CM, Bogers AJ, Piazza N, Kappetein AP. Aortic stenosis in the elderly: disease prevalence and number of candidates for transcatheter aortic valve replacement: a meta-analysis and modeling study. J Am Coll Cardiol. 2013 Sep 10;62(11):1002-12. doi: 10.1016/j.jacc.2013.05.015. Epub 2013 May 30. PMID 23727214
- [Background] Otto CM. Valvular aortic stenosis: disease severity and timing of intervention. J Am Coll Cardiol. 2006 Jun 6;47(11):2141-51. doi: 10.1016/j.jacc.2006.03.002. Epub 2006 May 15. PMID 16750677
- [Background] Carabello BA. Aortic stenosis: a fatal disease with but a single cure. JACC Cardiovasc Interv. 2008 Apr;1(2):127-8. doi: 10.1016/j.jcin.2007.12.004. No abstract available. PMID 19463289
- [Background] Vahanian A, Baumgartner H, Bax J, Butchart E, Dion R, Filippatos G, Flachskampf F, Hall R, Iung B, Kasprzak J, Nataf P, Tornos P, Torracca L, Wenink A; Task Force on the Management of Valvular Hearth Disease of the European Society of Cardiology; ESC Committee for Practice Guidelines. Guidelines on the management of valvular heart disease: The Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology. Eur Heart J. 2007 Jan;28(2):230-68. doi: 10.1093/eurheartj/ehl428. Epub 2007 Jan 26. No abstract available. PMID 17259184
- [Background] Gherli T, Colli A, Fragnito C, Nicolini F, Borrello B, Saccani S, D'Amico R, Beghi C. Comparing warfarin with aspirin after biological aortic valve replacement: a prospective study. Circulation. 2004 Aug 3;110(5):496-500. doi: 10.1161/01.cir.0000137122.95108.52. PMID 15289387
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811
- [Background] Attizzani GF, Ohno Y, Latib A, Petronio AS, Giannini C, Ettori F, Curello S, Bedogni F, Todaro D, Brambilla N, Bruschi G, Colombo P, Presbitero P, Fiorilli R, Poli A, Martina P, Colombo A, Barbanti M, Tamburino C. Acute and long-term (2-years) clinical outcomes of the CoreValve 31mm in large aortic annuli: A multicenter study. Int J Cardiol. 2017 Jan 15;227:543-549. doi: 10.1016/j.ijcard.2016.10.104. Epub 2016 Nov 1. PMID 27816304
- [Background] Nijhoff F, Agostoni P, Amrane H, Latib A, Testa L, Oreglia JA, De Marco F, Samim M, Bedogni F, Maisano F, Bruschi G, Colombo A, Van Boven AJ, Stella PR. Transcatheter aortic valve implantation in patients with severe aortic valve stenosis and large aortic annulus, using the self-expanding 31-mm Medtronic CoreValve prosthesis: first clinical experience. J Thorac Cardiovasc Surg. 2014 Aug;148(2):492-9.e1. doi: 10.1016/j.jtcvs.2013.09.059. Epub 2013 Nov 19. PMID 24263005
- [Background] Cilingiroglu M, Hakeem A. Fate of mitral regurgitation following transcatheter aortic valve implantation: the achilles heel of core valve? Catheter Cardiovasc Interv. 2011 Oct 1;78(4):645-6. doi: 10.1002/ccd.23359. No abstract available. PMID 21953759
- [Background] Bleiziffer S, Ruge H, Horer J, Hutter A, Geisbusch S, Brockmann G, Mazzitelli D, Bauernschmitt R, Lange R. Predictors for new-onset complete heart block after transcatheter aortic valve implantation. JACC Cardiovasc Interv. 2010 May;3(5):524-30. doi: 10.1016/j.jcin.2010.01.017. PMID 20488409